CLINICAL TRIAL: NCT05739539
Title: Assessment of Retinal Vascular Changes With and Without ILM Peeling in Diabetic Vitrectomy Using Optical Coherence Tomography Angiography.
Brief Title: Assessment of Retinal Vascular Changes With and Without ILM Peeling in Diabetic Vitrectomy Using OCT-A.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Essam Faseeh, Assistant Lecturer of Ophthalmology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1442022
Record Dates: First submitted 2023-01-27; First posted 2023-02-22 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Vitreous Hemorrhage; Tractional Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pars plana vitrectomy with ILM peeling (Active Comparator): Diabetic patients who fulfill the inclusion critera and will undergo pars plana vitrectomy and ILM peeling
  Interventions: Diagnostic Test: optical coherence tomography angiography; Diagnostic Test: spectral domain optical coherence tomography
- pars plana vitrectomy without ILM peeling (Active Comparator): Diabetic patients who fulfill the inclusion critera and will undergo pars plana vitrectomy without ILM peeling
  Interventions: Diagnostic Test: optical coherence tomography angiography; Diagnostic Test: spectral domain optical coherence tomography

INTERVENTIONS:
Diagnostic Test: optical coherence tomography angiography — optical coherence tomography angiography will be done postoperatively in both groups to assess the retinal microvascular changes
Diagnostic Test: spectral domain optical coherence tomography — optical coherence tomography for ganglion cell complex (GCC) measurement and assessment of macular edema or epiretinal membrane formation will be done postoperatively in both groups

SUMMARY:
Tractional retinal detachment (TRD) that involves the macula and non-clearing vitreous hemorrhage are the main causes of permanent vision loss in patients with diabetic retinopathy and requires prompt surgical intervention.

Macular peeling is a surgical technique used in many retinal diseases including diabetic retinal detachment.

Our purpose is to determine whether retinal microcirculatory changes occur after anatomically successful diabetic vitrectomy, and whether changes in blood flow vary if ILM peeling was done and whether changes in macular perfusion affect the final visual outcome.

The aim of this study is to non-invasively evaluate, with optical coherence tomography angiography (OCT-A), the anatomical changes of deep and superficial vascular density in the macula with and without macular peeling in diabetic vitrectomy.

DETAILED DESCRIPTION:
Background and Rationale:

Diabetic retinopathy (DR) is a leading cause of blindness among the working age group with increasing numbers of persons being affected worldwide.

The microvascular complications of diabetes result in macular leakage or exudation and vasoproliferative retinal disease, which are the hallmarks of advanced DR. Despite treatment of earlier stages of DR with medical therapy, several eyes will progress to require surgical treatment.

Surgical treatment for the advanced complications of DR can range from removal of a non-clearing vitreous hemorrhage, to more complicated surgical techniques such as in dealing with a combined tractional and rhegmatogenous retinal detachment (TRD/RRD) or tractional retinal detachment (TRD) involving or threatening the macula.

Tractional retinal detachment (TRD) that involves the macula is the main cause of permanent vision loss in patients with diabetic retinopathy and requires prompt surgical intervention. With the small-gauge vitrectomy system, anatomical success rate after pars plana vitrectomy (PPV) is reported to be over 90%.

Macular peeling is a surgical technique used in many retinal diseases including diabetic retinopathy, retinal detachment, macular holes, macular edema or foveal retinoschisis. The technique is based on surgical removal of the preretinal tissue or internal limiting membrane (ILM) in the macula.

PPV with ILM peeling has been reported to reduce retinal edema and improve visual acuity in patients with diabetic macula edema. However there is a controversial whether ILM peeling has benefit in patients undergoing PPV for PDR complications.

Studies found that fewer cases of epiretinal membranes and macular edema were observed postoperatively with ILM peeling in diabetic vitrectomy but visual acuity is similar with and without peeling.

In another recent study evaluating the benefits of ILM peeling in subjects undergoing PPV for the treatment of diabetic vitreous hemorrhage and found that better best-corrected visual acuity, fewer postoperative diabetic macular edema, and a lower incidence of epiretinal membrane at 6 months when ILM peeling was performed.

Optical coherence tomography angiography (OCTA) provides a non-invasive and quantitative approach for investigating retinal and choroidal microvasculature. The retinal vascular plexus of healthy subjects is formed by a superficial plexus located in the ganglion cell layer and nerve fiber layer, and a deep plexus located in the inner nuclear layers . The foveal capillary plexus forms a ring at the margin of the fovea, producing a capillary-free region called the foveal avascular zone (FAZ).

Our purpose is to determine whether retinal microcirculatory changes occur after anatomically successful diabetic vitrectomy, and whether changes in blood flow vary if ILM peeling was done and whether changes in macular perfusion affect the final visual outcome.

The aim of this study is to non-invasively evaluate, with optical coherence tomography angiography (OCT-A), the anatomical changes of deep and superficial vascular density in the macula with and without macular peeling in diabetic vitrectomy.

To our knowledge, there are presently no any studies evaluating OCT-A retinal vascular changes with and without ILM peeling after diabetic vitrectomy.

Objectives:

To assess the OCT-A retinal vascular changes with and without ILM peeling in diabetic vitrectomy patients.

- Methodology in details:

This prospective study will be conducted at Kasr Al-Aini Ophthalmology department and will include PDR patients who are candidates for PPV which will be recruited and assessed for eligibility for inclusion according to the above criteria.

All participants will be subjected to the following:

* Written informed consent.
* Detailed history including duration of diabetes, its treatment and glycemic control and systemic hypertension.
* History of ocular trauma, previous ocular surgery, history of treatment with intravitreal anti-VEGF or Argon retinal photocoagulation.
* Complete ophthalmic examination including best corrected visual acuity measurement, intraocular pressure, slit lamp examination and fundus examination.
* Pre-operative OCT-Angiography if possible in patients having clear media.
* Patients who are candidates for PPV will be assigned randomly using simple randomization with Microsoft Excel into one of two groups:

  * Group A: PPV with ILM peeling.
  * Group B: PPV without ILM peeling.
* 23-gauge PPV will be performed for patients in both groups , infusion pressure will be between 25-30 mmHg and in case of need to increase pressure for bleeding it will be less than 60 mmHg for no more than 5 minutes.
* Phacoemulsification & PCIOL will be done for cases with significant cataract.
* Silicone oil tamponade 1000 csk will be used for all cases. Follow up of the patients at 3 and 6 months after surgery with measuring BCVA, fundus examination, OCT-Angiography (optovue Inc) scan area of 3x3 mm and 6x6 mm to detect vascualr density: superficial capillary plexus (SCP), deep capillary plexus (DCP), foveal and parafoveal all quadrants using ETDRS circles, and the foveal avascular zone (FAZ) area and acirculatory index.
* OCT for measuring central macular thickness & ganglion cell complex (GCC) will be done.
* Patients' serial numbers only will be used on data collection sheets. Data will be entered on a computer with access limited to the researchers in order to ensure confidentiality of patients' information.

  * Intervention:
  * Therapeutic intervention (please describe):
  * Pars plana vitrectomy (PPV) will be performed for diabetic patients who meet the inclusion criteria, in group A: ILM peeling will be done and in group B: PPV without ILM peeling.
  * Diagnostic intervention (please describe):
  * OCT-A (optovue Inc) and OCT for measuring ganglion cell complex (GCC) will be done 3 and 6 months following surgery comparing both groups.
  * Does the research involve? Human participants
  * Type of consent of study participants:

Written consent

* Potential risks:

  * Iatrogenic Retinal break.
  * Infection.
  * Elevated intraocular pressure.
* Confidentiality of data:

None of the data obtained during the study will contain any personal information that can lead to patient identification, no personal photos for the patients will be obtained, no names or patients' identification numbers or records will be displayed.

Sample size (number of study subjects included and justification including the clinical and statistical assumptions supporting sample size calculation)

Total number of 36 eyes to be divided equally in 2 groups:

* Group A: 18 eyes will undergo PPV with ILM peeling.
* Group B: : 18 eyes will undergo PPV without ILM peeling.

Assuming equal number of eyes in two groups, power of study of 80%, statistical significance alpha of 0.05 (two sided). Based on data from literature [13] calculating minimal sample size needed to compare macular vascular density changes between two groups of diabetic vitrectomy with and without ILM peeling to detect difference of 3 % in vascular density with SD of 3 % using the following equation:

n= (2) (3) 2 (2.8) 2 / (3) 2 = 16 in each group

Assuming 10 % drop-out of cases the total number of cases will be 36 eyes.

Sampling technique: A convenient sample of patients with the inclusion and exclusion criteria will be assigned into study till reaching total sample size calculated.

Statistical analysis Data analysis packages will be SPSS version 21 Qualitative data will be presented by number and percentage , quantitative data will be presented by mean, standard deviation, median and interquartile range . Parametric and non-parametric tests of significant will be done chi square, Fisher exact for non-parametric data and student t test and ANOVA test for parametric data, man whitney test and mcnemar test for non parameteric data, Level of significance was set at p-value equal to or below 0.05.

Source of funding: (Please include source of funding even if self funding) Self funding

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old of both sexes.
* Patients having diabetic tractional retinal detachement threatening the macula (traction over posterior pole with attached fovea).
* Combined tractional-rhegmatogenous retinal detachement with attached macula.
* Diabetic persistent fibrovascular proliferation not responding to panretinal photocoagulation.
* Non clearing diabetic vitreous hemorrhage, subhyaloid hemorrhage.

Exclusion Criteria:

* Subject has had a previous vitrectomy (anterior or PPV) in the study eye.
* Subject has uncontrolled neovascular glaucoma (intraocular pressure > 30 mmHg despite medical/surgical treatment) in the study eye.
* Previous history of trauma in the study eye.
* Previous history of Anti-VEGF injection.
* Tractional macular detachment.
* Coexisting macular hole.
* Cases with previous arterial or venous occlusions.
* Coexisting posterior segment inflammation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Compare the superficial and deep vascular densities using OCT-A with and without ILM peeling in diabetic vitrectomy patients. | 18 months total study duration , 9 months follow up
  Compare the superficial and deep vascular densities in percentage compared to normative database using OCT-A (Optovue) with and without ILM peeling in diabetic vitrectomy patients.
Compare the foveal avascular zone using OCT-A between both groups. | 18 months total study duration , 9 months follow up
  Compare the foveal avascular zone measured in micrometer using OCT-A between both groups.

SECONDARY OUTCOMES:
Compare the best corrected visual acuity in both groups | 18 months total study duration , 9 months follow up
  Compare the best corrected visual acuity in both groups using decimal numbers on snellen's chart
Compare OCT ganglion cell complex (GCC) changes in both groups. | 18 months total study duration , 9 months follow up
  Compare OCT ganglion cell complex (GCC) changes in both groups measured as percentage of loss compared to age related normative database on the OCT device.
Compare incidence of epiretinal membrane formation in both groups. | 18 months total study duration , 9 months follow up
  Compare incidence of epiretinal membrane formation in both groups using OCT device either present or absent.
Compare incidence of macular edema in both groups. | 18 months total study duration , 9 months follow up
  Compare incidence of macular edema in both groups measured by calculating the central foveal thickness in micrometers using the OCT device

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Faseeh, MSc, Principal Investigator — KasrAlaini hospital
Locations (1):
- KasrAlaini hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No